CLINICAL TRIAL: NCT05987813
Title: A Pilot Study of Auricular Microstimulation to Determine if it Improves Vagal Modulation
Brief Title: Transcutaneous Electric Nerve Stimulation (TENS) for Vagal Modulation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: the ear clip is uncomfortable and compliance is down as a result. The team is working with manufacturer to develop new ear clip that will be used in a new protocol.
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM20025635
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Functional Gastrointestinal Disorders
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Intervention Model Description: FGID group, non-FGID group. Assigned to 2 hours of daily TENS usage
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- FGID (Experimental): Patients with a FGID
  Interventions: Device: TENS Unit
- Non-FGID (Experimental): Patients without a FGID
  Interventions: Device: TENS Unit

INTERVENTIONS:
Device: TENS Unit — Usage of the Transcutaneous Electrical Nerve Stimulation device for 2 hours a day.

SUMMARY:
This study is to determine if the auricular microstimulator produces the expected increase in HRV.

DETAILED DESCRIPTION:
The aim of this proposal is to determine if utilizing an affordable tool like microstimulation utilizing a transcutaneous electric nerve stimulator (TENS) unit and applying the stimulation to the ear though an ear clip does improve vagal modulation. This can be easily done at home by utilizing the microstimulation for 2 hours/day and measuring vagal modulation before and after. Previous research investigating this had participants use the unit for 2 hours as well (Chelimsky et al., 2019), however the data from this study was inconclusive, and therefore this study aims to demonstrate effectiveness of the unit usage on heart rate variability (HRV).

Although functional gastrointestinal disorders (FGID) affect 10%-20% of children and adolescents. 1-3 the pathophysiology remains unknown. The multiple current hypotheses include visceral hypersensitivity, altered brain-gut connections, dysbiosis, genetic and epigenetic factors, and increased gut permeability among others. 4 Since the vagus nerve links the brain to the gut, many studies of adult subjects have evaluated the cardiovagal modulation in this group of disorders. The cardiovagal modulation can be measured by heart rate variability (HRV). HRV evaluates the heart rate fluctuation over a period of time. HRV is considered a reliable tool to look at parasympathetic function, baroreflex function, and parasympathetic to sympathetic balance.5, 6 High-frequency (hf) HRV is a marker of vagal modulation. The low-frequency (lf) HRV probably reflects cardiac autonomic outflow from the baroreflex or parasympathetic regulation, rather than sympathetic modulation, although this is still being discussed.6, 7

A meta-analysis of adult subjects with irritable bowel syndrome (IBS) showed decreased cardiovagal modulation.8 One study compared children aged 7-10 years of age with functional abdominal pain or IBS to healthy subjects. They found no difference in cardiovagal and cardiac sympathetic modulation.9 However, a study of young adolescents with different chronic pain syndromes, including chronic abdominal pain, showed decreased cardiovagal modulation.10 These findings are similar to those in many adult syndromes with chronic pain, such as chronic pelvic pain,11 complex regional pain syndrome,12 fibromyalgia,13 and chronic neck pain.14

Although future research would aim to investigate vagal modulation in those specifically with FGID, for preliminary data purposes we are testing the unit's effects on heart rate variability regardless of having/not having an FGID diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 12 - 21 years old
* Either diagnosed OR not diagnosed with chronic idiopathic nausea, functional abdominal pain, dyspepsia and/or irritable bowel syndrome.
* English speaking

Exclusion Criteria:

* Patients who are unable to stand upright during the heart rate variability recording
* Patients with a known bleeding disorder
* Patients with swollen, infected, inflamed, or other skin eruptions on outer ear
* Patients with epilepsy
* Patients with any implanted cardiac pacemaker or defibrillator
* Patients with serious arterial circulatory problems in the lower limbs
* Patients with abdominal or inguinal hernia
* Patients who are pregnant
* Any unstable medical condition, such as renal disease, uncontrolled diabetes, etc.
* Requires new medication during the 4 weeks of the study that may affect the gastrointestinal symptoms, vagal modulation or immune response.
* Practices over 1 hour of aerobic activity a day
* Daily practice of abdominal breathing (yoga)

Ages: 12 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2023-10-18 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gisela Chelimsky, MD, Principal Investigator — VCU
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Anonymized information may be shared to other researchers for future relevant projects.

REFERENCES:
- [Background] Hyams JS, Davis P, Sylvester FA, Zeiter DK, Justinich CJ, Lerer T. Dyspepsia in children and adolescents: a prospective study. J Pediatr Gastroenterol Nutr. 2000 Apr;30(4):413-8. doi: 10.1097/00005176-200004000-00012. PMID 10776953
- [Background] APLEY J, NAISH N. Recurrent abdominal pains: a field survey of 1,000 school children. Arch Dis Child. 1958 Apr;33(168):165-70. doi: 10.1136/adc.33.168.165. No abstract available. PMID 13534750
- [Background] Boey C, Yap S, Goh KL. The prevalence of recurrent abdominal pain in 11- to 16-year-old Malaysian schoolchildren. J Paediatr Child Health. 2000 Apr;36(2):114-6. doi: 10.1046/j.1440-1754.2000.00465.x. PMID 10760006
- [Background] Enck P, Aziz Q, Barbara G, Farmer AD, Fukudo S, Mayer EA, Niesler B, Quigley EM, Rajilic-Stojanovic M, Schemann M, Schwille-Kiuntke J, Simren M, Zipfel S, Spiller RC. Irritable bowel syndrome. Nat Rev Dis Primers. 2016 Mar 24;2:16014. doi: 10.1038/nrdp.2016.14. PMID 27159638
- [Background] Riganello F, Garbarino S, Sannita WG. Heart Rate Variability, Homeostasis, and Brain Function. J Psychophysiol. 2012; 26: 178- 203.
- [Background] Goldstein DS, Bentho O, Park MY, Sharabi Y. Low-frequency power of heart rate variability is not a measure of cardiac sympathetic tone but may be a measure of modulation of cardiac autonomic outflows by baroreflexes. Exp Physiol. 2011 Dec;96(12):1255-61. doi: 10.1113/expphysiol.2010.056259. Epub 2011 Sep 2. PMID 21890520
- [Background] Reyes del Paso GA, Langewitz W, Mulder LJ, van Roon A, Duschek S. The utility of low frequency heart rate variability as an index of sympathetic cardiac tone: a review with emphasis on a reanalysis of previous studies. Psychophysiology. 2013 May;50(5):477-87. doi: 10.1111/psyp.12027. Epub 2013 Feb 27. PMID 23445494
- [Background] Liu Q, Wang EM, Yan XJ, Chen SL. Autonomic functioning in irritable bowel syndrome measured by heart rate variability: a meta-analysis. J Dig Dis. 2013 Dec;14(12):638-46. doi: 10.1111/1751-2980.12092. PMID 23927739
- [Background] Jarrett M, Heitkemper M, Czyzewski D, Zeltzer L, Shulman RJ. Autonomic nervous system function in young children with functional abdominal pain or irritable bowel syndrome. J Pain. 2012 May;13(5):477-84. doi: 10.1016/j.jpain.2012.02.007. Epub 2012 Apr 20. PMID 22520688
- [Background] Evans S, Seidman LC, Tsao JC, Lung KC, Zeltzer LK, Naliboff BD. Heart rate variability as a biomarker for autonomic nervous system response differences between children with chronic pain and healthy control children. J Pain Res. 2013 Jun 12;6:449-57. doi: 10.2147/JPR.S43849. Print 2013. PMID 23788839
- [Background] Williams DP, Chelimsky G, McCabe NP, Koenig J, Singh P, Janata J, Thayer JF, Buffington CA, Chelimsky T. Effects of Chronic Pelvic Pain on Heart Rate Variability in Women. J Urol. 2015 Nov;194(5):1289-94. doi: 10.1016/j.juro.2015.04.101. Epub 2015 May 9. PMID 25963185
- [Background] Mork PJ, Nilsson J, Loras HW, Riva R, Lundberg U, Westgaard RH. Heart rate variability in fibromyalgia patients and healthy controls during non-REM and REM sleep: a case-control study. Scand J Rheumatol. 2013;42(6):505-8. doi: 10.3109/03009742.2012.755564. Epub 2013 Feb 20. PMID 23425526
- [Background] Terkelsen AJ, Molgaard H, Hansen J, Finnerup NB, Kroner K, Jensen TS. Heart rate variability in complex regional pain syndrome during rest and mental and orthostatic stress. Anesthesiology. 2012 Jan;116(1):133-46. doi: 10.1097/ALN.0b013e31823bbfb0. PMID 22089824
- [Background] Kang JH, Chen HS, Chen SC, Jaw FS. Disability in patients with chronic neck pain: heart rate variability analysis and cluster analysis. Clin J Pain. 2012 Nov-Dec;28(9):797-803. doi: 10.1097/AJP.0b013e3182442afd. PMID 22751023
- [Background] Chelimsky G, Rausch S, Bierer D, Feng M, Simpson P, Awe E, Chelimsky T. Cardiovagal modulation in pediatric functional gastrointestinal disorders. Neurogastroenterol Motil. 2019 May;31(5):e13564. doi: 10.1111/nmo.13564. Epub 2019 Mar 27. PMID 30916860

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FGID | Non-FGID
Started | 5 | 3
Completed | 5 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FGID | Non-FGID | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 0 | 5
  Between 18 and 65 years | 0 | 3 | 3
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 17 (0.707) | 19 (0) | 17.75 (1.165)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in High-frequency Heart Rate Variability (hfHRV) at 4 Weeks
Description: Determine if microstimulation over a 4 week period results in improvement in hfHRV power.
  Average hfHRV power was calculated at baseline and 4 weeks. The change in average hfHRV power in milliseconds squared from baseline to 4 weeks was calculated for each participant. The average change for each group is reported.
Time Frame: Assessed at baseline and 4 weeks.
Measure: Mean (Standard Deviation); unit: ms squared
Arm/Group | FGID | Non-FGID
Number analyzed (Participants) | 5 | 3
ms squared | 23.517 (31.705) | 11.69 (19.644)

2. Primary Outcome: Rate of Compliance With Daily TENS Usage
Description: Determine the compliance rate of adolescents utilizing a microstimulator.
  Compliance rate calculated as number of minutes unit was used (summed from all self-report daily recording journals) divided by 3360 (the total number of minutes the unit could have been used if the participant used it for 2 hours daily for 4 weeks). The rate average for each group is reported.
Time Frame: Assessed daily for duration of study (4 weeks) via self-report recording journal.
Measure: Mean (Standard Deviation); unit: percentage - compliance rate
Arm/Group | FGID | Non-FGID
Number analyzed (Participants) | 5 | 3
percentage - compliance rate | 0.598 (0.296) | 0.823 (0.211)

ADVERSE EVENTS:
Time Frame: Duration of study participation- 4 weeks
Description: Participants could report AEs in a section of their Daily Recording Diary, completed virtually each day via REDCap data capture system.
Arm/Group | FGID | Non-FGID
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/3
Other Adverse Events (participants affected / at risk) | 4/5 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FGID (N=5) | Non-FGID (N=3)
Ear clip discomfort (Ear and labyrinth disorders) | 4 (8) | 3 (3) — Participants reported ear discomfort while wearing TENS unit ear clips.
Ear scabbing (Ear and labyrinth disorders) | 3 (7) | 0 (0) — Participants reported mild scabbing as a result of wearing the TENS unit ear clips daily.
Blurry vision (Eye disorders) | 1 (1) | 0 (0) — Participant reported blurry vision that spontaneously resolved later the same day.
Headache (General disorders) | 1 (1) | 0 (0) — Participant reported a headache one day after using the unit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-04-23): https://cdn.clinicaltrials.gov/large-docs/13/NCT05987813/Prot_002.pdf
  • Informed Consent Form (2024-06-26): https://cdn.clinicaltrials.gov/large-docs/13/NCT05987813/ICF_001.pdf